CLINICAL TRIAL: NCT06013228
Title: Trajectories of Fatigue, Glycated Hemoglobin, Diabetes Self-management, and Quality of Life in People With a Dual Diagnosis of Operable Pancreatic Tumor and Diabetes Mellitus: A Longitudinal Mixed-methods Study
Brief Title: Trajectories of Fatigue and Quality of Life in People With Both Operable Pancreatic Tumor and Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202302123RIND
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-08

CONDITIONS: Operable Pancreatic Tumor; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In people with both burdens of OPT and DM, fatigue is the most common and deliberating symptom that likely impacts their quality of life and diabetes self-management. However, little is known about the longitudinal relationships among fatigue, its influencing factors, glycemic status, diabetes self-management, and quality of life in people with both OPT and DM during the first-year post-operation. Thus, the purposes of this study are to (1) describe the trajectories of fatigue, HbA1c, diabetes self-management, and quality of life in people with OPT and DM within 12 months post-operation; (2) examine the relationships among the trajectories of fatigue, its influencing factors, diabetes self-management, and quality of life in people with OPT and DM; and (3) understand the experiences of people with both OPT and DM regarding changes in challenges with diabetes, fatigue, diabetes self-management, diabetes care needs, and quality of life.

DETAILED DESCRIPTION:
Pancreatic cancer is a devastating disease, and surgery is one of the treatment options with the goal of curing the disease. However, people with operable pancreatic tumor (OPT) often have a high prevalence of comorbid diabetes mellitus (DM) that is likely to result in increased glucose fluctuation and poor glycemic control. Importantly, in people with both burdens of OPT and DM, fatigue is the most common and deliberating symptom that likely impacts their quality of life and diabetes self-management. However, little is known about the longitudinal relationships among fatigue, its influencing factors, glycemic status, diabetes self-management, and quality of life in people with both OPT and DM for 12 months of follow-up. Thus, the purposes of this study are to (1) describe the trajectories of fatigue, HbA1c, diabetes self-management, and quality of life in people with OPT and DM within 12 months of follow-up; (2) examine the relationships among the trajectories of fatigue, its influencing factors, diabetes self-management, and quality of life in people with OPT and DM; and (3) understand the experiences of people with both OPT and DM regarding changes in challenges with diabetes, fatigue, diabetes self-management, diabetes care needs, and quality of life. Guided by the Theory of unpleasant symptoms, this two-year study will use a longitudinal concurrent mixed methods design. Participants will be recruited from an outpatient pancreatic surgical department at a medical center in northern Taiwan using purposive sampling. For the quantitative component, data will be collected using structured questionnaires over five time points (baseline, 3, 6, 9, and 12 months post baseline),The Chinese version of a structured questionnaire, including the demographic and clinical characteristics form, Diabetes Distress Scale, Center for Epidemiological Studies Depression Scale, Multidimensional Scale of Perceived Social Support, Fatigue Symptom Inventory, Summary of Diabetes Self-Care Activities, and the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire will be used. For data analysis, latent growth curve modeling under a structural equation modeling framework using Mplus version 8.6 will be performed. A sample of 115 participants with both OPT and DM will be recruited. To illuminate our understanding of the findings from the quantitative component of the study, the qualitative component will use semi-structured qualitative interviews to explore the changes in challenges with diabetes, fatigue, diabetes self-management, diabetes care needs, and quality of life for a subsample of 20 participants who reported their fatigue intensity scores as 4 or more on the Fatigue Symptom Inventory concurrently. Qualitative content analysis will be used to analyze the qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Operable pancreatic tumor within 5 years and are following up at the outpatient department
* Diagnosed with diabetes mellitus
* Aged 18 or above
* Can communicate in Mandarin or Taiwanese
* Agree to participate and sign the informed consent form

Exclusion Criteria:

* Under active treatment for cancer other than pancreatic tumor
* Have a cognitive impairment
* Do not know that they have pancreatic tumor
* Diagnosed with chronic fatigue syndrome or fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from a pancreatic surgical outpatient department (OPD) at a medical center located in northern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | baseline, 3, 6, 9, and 12 months post baseline
  Fatigue Symptom Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Ju Kuo, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will only be available to other researchers on reasonable request and only de-identified data will potentially be available to protect the rights of the participants.